CLINICAL TRIAL: NCT03181035
Title: Defining a Personalized Hypoxic Radiation Target Through Correlation of Functional F18-FAZA PET Imaging to Pimonidazole-stained 3D Whole-mounted Histological Specimen
Brief Title: Correlation of FAZA PET Hypoxia Imaging To 3D Histology in Oral Tongue Cancer
Acronym: FAITH
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Pause to enrolment due to COVID-19 pandemic and protocol amendment (change to equipment used)
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAITH 253-2015; NCT02519959 (obsolete NCT alias)
Record Dates: First submitted 2017-04-17; First posted 2017-06-08 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Tongue Cancer
Keywords: Oral Tongue Cancer; Tumor Hypoxia
MeSH Terms: conditions — Tongue Neoplasms | interventions — pimonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAZA and pimonidazole (Experimental): (18)F-Fluoroazomycin arabinoside (FAZA) will be administered via intravenous injection at a dose of 5.2 MBq/kg with a minimum dose of 200 Megabecquerel (MBq) (5.4 Millicurie (mCi)) and a maximum dose of 600 MBq (16.2 mCi) prior to positron emission tomography (PET) imaging. A single dose of oral pimonidazole capsules at a dose of 0.5 g/m2, will be taken by participants 16-20 hours prior to tumor resection surgery.
  Interventions: Radiation: (18)F-Fluoroazomycin arabinoside; Drug: Pimonidazole

INTERVENTIONS:
Radiation: (18)F-Fluoroazomycin arabinoside — FAZA PET diagnostic testing
  Other Names: FAZA
Drug: Pimonidazole — oral pimonidazole hypoxia labeling

SUMMARY:
This is a pilot study in the form of a prospective Phase II, single centre, single arm hypoxia study of oral tongue cancer with FAZA-PET imaging and pimonidazole targeted IHC of surgical specimens.

DETAILED DESCRIPTION:
In head and neck cancer, areas of tumours with low oxygen supply (called tumour hypoxia) harbour cells that are resistant to radiation and are prone to metastasize. Modern radiotherapy techniques are precise enough to deliver radiation to these small areas and could be used to target these areas to receive higher doses of radiation than the rest of the tumour to overcome resistance. Hypoxia can be "seen" in the body using special imaging such as [F-18]-FAZA-PET ([F-18]-Fluoroazomycin arabinoside positron emission tomography) but it has not been tested as a method for creating radiation treatment targets. As part of regular pathology tumour tissue is sliced extremely thinly (<1/100th of a millimeter) and stained so that individual cells can be seen under a microscope. Immunohistochemistry (IHC) is a special type of "stain" that can specifically highlight hypoxic areas. This method is considered the most accurate way to inspect for the presence of hypoxia. There is not a specific staining target for hypoxia ordinarily, but when patients ingest a substance called pimonidazole hydrochloride (HCl) it builds up specifically in hypoxic areas and can be targeted for IHC staining. In this study participants with oral tongue cancer will have a [F-18]-FAZA-PET scan and take a single dose of oral pimonidazole-HCl before having surgery to remove their cancer. The whole tumour will be used to create microscope slides using very thin slices of the tumour. The slices will be stained using IHC to show where the pimonidazole has built up and digital scans of the slides will be made. The hypoxia seen on the FAZA-PET scan will be "matched" with hypoxia on the electronic slides to see if the FAZA truly shows where hypoxia is in tumours and if it could be used as a way to plan radiation treatments to deliver more radiation to just those areas.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Stage II-III oral tongue squamous cell carcinoma
* Naïve to treatment for resectable disease
* Surgical resection as definitive treatment modality
* Ability to participate and willingness to give written informed consent prior to performance of any study-related procedures and to comply with the study protocol
* Adequate hematologic, renal and liver function as defined by the following laboratory values up to 30 days prior to commencement of dosing (administration of FAZA):

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 50 ×109/L
  * Hemoglobin ≥ 9 g/dL
  * Bilirubin ≤ 1.5 × upper limit of normal (ULN) (20.0 µmol)
  * Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5 × the ULN (37 U/L, 40 U/L, 120 U/L)
  * Serum creatinine ≤ 1.5 × the ULN (106 µmol/L) or creatinine clearance ≥ 50 mL/min on the basis of the Cockroft-Gault glomerular filtration rate estimation: [(140-age) × (weight in kg × (0.85 if female)]/[72 × (serum creatinine in mg/dL)]
  * Prothrombin time (PT), international normalized ratio (INR), partial thromboblastin time (PTT) ≤ 1.5 × the ULN (respectively 1.1, 14 sec, 35 sec)
* Negative serum pregnancy test within 14 days prior to commencement of dosing in women of childbearing potential. Women of non-childbearing potential need not undergo pregnancy testing. Female participants of childbearing potential agree to use adequate methods of contraception from the time of enrollment until 28 days after surgery. Clinically acceptable methods of birth control for this study include intrauterine devices (IUD), birth control pills, hormonal implants, injectable contraceptives, and using barrier methods such as condoms, vaginal diaphragm with spermicide, or sponge.

Exclusion Criteria:

* Patients who have received prior chemotherapy or radiation therapy for their oral tongue carcinoma
* Stage I, Stage III T1/N1/M0, and Stage IV disease
* Pregnant or breastfeeding at the time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cellular hypoxia correlation | 1 year
  The degree to which hypoxic signal measured by FAZA-PET imaging is correlated with true cellular hypoxia confirmed by immunohistochemical staining of pimonidazole using a 3D whole-mount approach
Hypoxic reference standard | 1 year
  A reference standard hypoxic radiation target will be defined through the correlation of functional F18-FAZA PET imaging to a pimonidazole-stained 3D whole mounted histological specimen.

SECONDARY OUTCOMES:
Registration quality | 1 year
  The quality of registration will be assessed through measuring registration error of various automatic and semi-automatic co-registration techniques
Textural feature comparison | 1 year
  Potential relationships between textural features of MRI, PET-CT, and immunohistochemistry will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Poon, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided